CLINICAL TRIAL: NCT03727113
Title: Optimization of Antibiotic Treatment in Hematopoietic Stem Cell Receptors: Impact on Intestinal Microbiota and in Clinical Outcomes
Brief Title: Optimization of Antibiotic Treatment in Hematopoietic Stem Cell Receptors
Acronym: Optimbioma
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: Optimbioma
Record Dates: First submitted 2018-10-16; First posted 2018-11-01 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Hematopoietic Stem Cell Transplantation; Graft Versus Host Disease
Keywords: microbiota; microbiome; graft versus host disease; infection; antibiotics
MeSH Terms: conditions — Graft vs Host Disease; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control cohort: Patients receiving an allogeneic hemopoietic stem cell transplant in Centers using a classical strategy of administration of antibiotics.
  Interventions: Procedure: Control cohort
- Optimization cohort: Patients receiving an allogeneic hemopoietic stem cell transplant in Centers using an optimization/antibiotic strategy.
  Interventions: Procedure: Optimization cohort

INTERVENTIONS:
Procedure: Optimization cohort — Recipients of an allogeneic hemopoietic stem cell transplant in Centers using an optimization/antibiotic strategy.
  Groups: Optimization cohort
Procedure: Control cohort — Recipients of an allogeneic hemopoietic stem cell transplant in Centers using a classical strategy of administration of antibiotics.
  Groups: Control cohort

SUMMARY:
There are data suggesting that the reduction of the diversity of intestinal microbiota caused by the used treatments in the setting of allogeneic hemopoietic stem cell transplant (ASCT), and specially antibiotics, may be related to increased incidence of graft versus host disease (GVHD) and worst clinical outcomes. Present "European Conference on Infections in Leukaemia" guidelines exhort to antibiotic treatment optimization in hematological patients, without excluding ASCT receptors. This study aims to demonstrate that in ASCT receptors a predefined protocol of optimization of the antibacterial treatment will preserve the intestinal microbiota diversity which will correlate with decrease incidence of acute GVHD. And that this procedure is safe because it will not worsen the incidence of infections, transplant related mortality, infectious mortality or global survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to receive their first allogeneic hematopoietic transplant as a treatment of any disease.
* Conformity of the patient to participate by signing the informed consent.
* Patients who have received a previous autologous transplant are not excluded.

Exclusion Criteria:

* Non-compliance of the patient to sign the informed consent.
* Patients who have already started the conditioning (or thereafter) will not be included.
* Allograft recipients who have previously received the transplant will not be included. Second allogeneic transplants are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (> 18 years old) who are going to receive their first hematopoietic allogeneic transplant of any modality and who sign the informed consent to participate in this study will be included.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Impact on microbiota | From the Previous Day of starting conditioning treatment until the last documented day of antibiotherapy or hospital discharge, whichever came first, assessed up to one month post-transplant.
  Comparison of biological alpha and beta diversity of the intestinal microbiota of both study groups (classical and optimized antibiotherapy). Calculation of alpha diversity (OTUs richness and Shannon diversity indexes observed, Faith's Phylogenetic Diversity and Evenness) and beta diversity (Jaccard distance, Bray-Curtis distance, Unweighted UniFra distance, used for comparing biological communities) indexes by QIIME 2 (microbiome bioinformatics platform).

SECONDARY OUTCOMES:
Incidence of Acute graft versus host disease | From the day of transplant (Day 0) to Day +100 posttransplant
  Comparison of the incidence of any degree, degree-II and degree-III/IV of acute graft versus host disease between the groups of patients with high and low diversity in their microbiota. Cumulative Incidence curve estimation.
  Test for the comparison of groups: Gray Test.
Transplant related mortality | From the day of transplant (Day 0) to Days +30, +100 and +365 posttransplant
  Comparison of transplant related mortality between both study groups (classical and optimized antibiotherapy). Cumulative Incidence curve estimation. Test for the comparison of groups: Gray Test.
Mortality caused by infection | From the day of transplant (Day 0) to Days +30, +100 and +365 posttransplant
  Comparison of infection related mortality between both study groups (classical and optimized antibiotherapy. Cumulative Incidence curve estimation. Test for the comparison of groups: Gray Test.
Incidence of severe infections | From the day of transplant (Day 0) to Day +30 posttransplant
  Comparison of the incidence of severe infections between both study groups (classical and optimized antibiotherapy). Cumulative Incidence curve estimation. Test for the comparison of groups: Gray Test.
Overall survival | From the day of transplant (Day 0) to Days +30, +100 and +365 posttransplant
  Comparison of overall survival between both study groups (classical and optimized antibiotherapy) Kaplan-Meier curve estimation. Test for the comparison of groups: Log-Rank Test.
Disease free survival | From the day of transplant (Day 0) to Days +30, +100 and +365 posttransplant
  Comparison of the diseae free survival between both study groups (classical and optimized antibiotherapy Kaplan-Meier curve estimation. Test for the comparison of groups: Log-Rank Test.

CONTACTS AND LOCATIONS:
Overall Officials: Ildefonso Espigado, PhD, MD, Principal Investigator — Hematology Service, Hematopoietic Transplant Program, Seville Biomedicine Institute (IBIS) - Virgen del Rocío University Hospital, Seville.
Locations (5):
- Spain (5):
  - Virgen del Rocío University Hospital, Seville., Seville, Seville
  - Gregorio Marañón University Hospital, Madrid
  - Salamanca University Hospital, Salamanca
  - Marqués de Valdecilla University Hospital, Santander
  - University Clinical Hospital of Valencia, Valencia

REFERENCES:
- [Background] Aguilar-Guisado M, Espigado I, Martin-Pena A, Gudiol C, Royo-Cebrecos C, Falantes J, Vazquez-Lopez L, Montero MI, Rosso-Fernandez C, de la Luz Martino M, Parody R, Gonzalez-Campos J, Garzon-Lopez S, Calderon-Cabrera C, Barba P, Rodriguez N, Rovira M, Montero-Mateos E, Carratala J, Perez-Simon JA, Cisneros JM. Optimisation of empirical antimicrobial therapy in patients with haematological malignancies and febrile neutropenia (How Long study): an open-label, randomised, controlled phase 4 trial. Lancet Haematol. 2017 Dec;4(12):e573-e583. doi: 10.1016/S2352-3026(17)30211-9. Epub 2017 Nov 15. PMID 29153975
- [Background] Averbuch D, Orasch C, Cordonnier C, Livermore DM, Mikulska M, Viscoli C, Gyssens IC, Kern WV, Klyasova G, Marchetti O, Engelhard D, Akova M; ECIL4, a joint venture of EBMT, EORTC, ICHS, ESGICH/ESCMID and ELN. European guidelines for empirical antibacterial therapy for febrile neutropenic patients in the era of growing resistance: summary of the 2011 4th European Conference on Infections in Leukemia. Haematologica. 2013 Dec;98(12):1826-35. doi: 10.3324/haematol.2013.091025. PMID 24323983
- [Derived] Jimenez-Jorge S, Labrador-Herrera G, Rosso-Fernandez CM, Rodriguez-Torres N, Pachon-Ibanez ME, Smani Y, Marquez-Malaver FJ, Limon Ramos C, Solano C, Vazquez-Lopez L, Kwon M, Mora Barrios JM, Aguilar-Guisado M, Espigado I; GETH (Grupo Espanol de Trasplante Hematopoyetico y Terapia Celular). Assessing the impact on intestinal microbiome and clinical outcomes of antibiotherapy optimisation strategies in haematopoietic stem cell transplant recipients: study protocol for the prospective multicentre OptimBioma study. BMJ Open. 2020 Jul 20;10(7):e034570. doi: 10.1136/bmjopen-2019-034570. PMID 32690735